CLINICAL TRIAL: NCT03401060
Title: Interest of Denosumab Treatment in Osteoporosis Associated to Systemic Mastocytosis
Acronym: DenosuMast
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CEREMAST (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P150918J; 2016-000596-25 (EudraCT Number)
Record Dates: First submitted 2018-01-04; First posted 2018-01-17 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis; Systemic Mastocytosis
Keywords: Systemic mastocytosis; Osteoporosis; Bone mineral density (BMD); Denosumab; RANKL
MeSH Terms: conditions — Osteoporosis; Mastocytosis, Systemic | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental medication 1 (Experimental): Denosumab 60 mg subcutaneously injection with prefilled syringe
  Interventions: Drug: Denosumab
- Experimental medication 2 (Placebo Comparator): NaCl 0.9%, 20ml phial, solution for injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab — Each subcutaneous injection will occur every 6 months during 3 years for a total of 7 injections
  Other Names: XGeva®
  Arms: Experimental medication 1
Drug: Placebo — Each subcutaneous injection will occur every 6 months during 3 years for a total of 7 injections
  Arms: Experimental medication 2

SUMMARY:
The study is looking at the efficacy of subcutaneously administrated denosumab 60 mg every 6 months versus placebo after 3 years, by analyze of lumbar spine bone mineral density (BMD) in systemic mastocytosis.

Investigators hypothesize that use of denosumab subcutaneously in patients with osteoporosis related to systemic mastocytosis is effective and safe to improve bone mineral density and prevent new bone events, based on targeted specific RANKL secretion by mast cells and short half-life of denosumab.

DETAILED DESCRIPTION:
Systemic mastocytosis (SM) represents a heterogenous group of disease characterized by abnormal proliferation of mast cells caused by activating mutations in c-Kit receptor; a tyrosine kinase family receptor present in mast cell that control cell proliferation. Prevalence of SM is estimated to 1/20 000 person. According to the World Health Organization (WHO) criteria (Johnson et al, 2009), SM can be separated into two different groups : indolent SM and aggressive SM.

Aggressive SM are defined by a poor prognostic disease either because of an important mast cell tumor mass as sarcoma mastocytosis or mast cell leukemia, or due to an association with an other myeloid hemopathy as myelodysplasic/myeloproliferative syndrome.

Indolent SM are the most common cases with a very good prognostic similar to general population. Symptoms related to mast cell proliferation in indolent SM are very various (Theoharides et al., 2015) and could be divided into 2 entities : those related to mast cell proliferation in tissue as the urticaria pigmentosa and those related to the mast cell degranulation.

There are many clinical relevant mediators released by mast cells after activation that could have putative effects on different systems as cardiovascular, cutaneous, neurologic, digestive, systemic, respiratory and musculoskeletal (Frenzel et al., 2013). Tryptase, histamine, prostaglandin, interleukine-6 and Tumor Necrosis Factor (TNF)-α are the most common and ubiquitous mediators released by mast cells but there are also some specific mediator targeting an organ as RANKL ; expression of RANKL by mast cells directly control regulation of osteoclast activity and is involved in osteoporosis associated to SM (Rabenhorst et al., 2013).

In systemic mastocytoses, bone lesions are found in about half of patients. A third have osteoporosis defined as a lumbar spine or hip bone T score of -2,5 Standard Deviation (SD) or less. In most cases, osteoporosis was complicated at least by one vertebral fracture with pain and functional disorders (Barete et al, 2010). The median time to fragility fracture after mastocytoses diagnosis is up to 5 years, even in very young population usually considering as low risk of fracture in non mastocytoses associated osteoporosis (Van de Veer et al., 2014)

By default, these patients are generally treated with bisphosphonate per os or intravenously with some efficiency on bone mineral density gain and bone turnover marker decrease (Rossini et al, 2014). However, no study with bisphosphonate in SM has showed durable prevention of new bone events and there are no randomized studies that proved their efficacy in systemic mastocytosis. Moreover, these drugs are not well tolerated in SM wether per os due to worsening of digestive symptoms by mast cells activation, or intravenously with an important number of acute phase characterized by some systemic symptoms as fever ; really experiences with intravenous biphosphonate but very increased in SM. Additional, the use of a bisphosphonate ask the question of the residual long-term effect of this drug that may be several years or even decades with a significant risk of atypical fracture secondary to a adynamic bone remodeling (Edwards et al. , 2013) and the long-term presence of crystals of bisphosphonate in the skeleton, particularly worrying in women of childbearing age. In postmenopausal osteoporosis, importance of residual long-term effect is weighted with advanced median age of patient. The fact that mostly patients with a systemic mastocytosis are young people led to restrict the use of bisphosphonate due to those effects.

Among different treatment available in post menopausal osteoporosis, the use of an anti-RANKL antibody, denosumab, in SM associated osteoporosis could be interesting. First, denosumab has already shown significant efficacy in the treatment of postmenopausal osteoporosis in women (Cummings et al , 2009). Second, this treatment is proposed every 6 months by a subcutaneous injection with very few side effects and half-life drug is shorter than biphosphonate with probably low residual long-time effect. Third, as mast cells expressed mainly RANKL with a direct role on bone turnover in SM. The use of a specific drug seems to be obvious and attractive.

ELIGIBILITY:
Inclusion Criteria:

* Male or female >/= 18 years of age at time of informed consent
* Willingness and ability to sign informed consent, comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
* Patient with Indolent systemic or cutaneous mastocytosis according to WHO criteria (Appendix 4) with any specific treatment including corticosteroid, chemotherapy and immunomodulating drugs.
* Patient with:

  * osteoporosis defined as bone mineral density T score ≤ -2.5 at the lumbar spine, OR
  * osteopenia defined as BMD T-score >-2,5 and ≤ -1 at the lumbar spine and low energy fracture (defined as fractures that are associated with decreased bone mineral density. Are excluded fractures of skull, face, mandible, metacarpals, fingers, or toes, pathologic fracture, and fracture that are associated with severe trauma).

(in case of osteoarthritis at the lumbar spine, the T score at left femoral neck or total left hip can be used to define osteoporosis or osteopenia)

Exclusion Criteria:

* Patient with aggressive mastocytosis or/and Associated Hematologic Non-Mastocytosis Disease (AHNMD)
* Patient with conditions that influence bone metabolism (primitive hyperparathyroidism, hyperaldosteronism, hypercorticism, etc …)
* Patient treated with intravenous bisphosphonate within 1 year prior to enrolment or with any other antiosteoporotic treatment within 3 months before enrolment. (per os bisphosphonate, strontium ranelate) Calcium and vitamin supplementation will be accepted
* Patient previously treated with denosumab
* Patient with hypocalcemia and/or hypo25-hydroxyvitamin D level non substituted prior enrolment
* Woman without contraceptive treatment if of childbearing age.
* Pregnant or breastfeeding woman
* Patient with contraindication to denosumab
* Patient with medical, psychiatric or other conditions that may interfere with patient safety
* Patient with dental problem that need any dental surgery within 6 months after enrolment.
* Patient with clearance of creatinine less than 30 mL/min/1,73m2 (MDRD) or patient receiving dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Analysis of the lumbar spine bone mineral density (BMD) | 3 years
  Dual energy x-ray absorptiometry at lumbar spine (L2-L4)

SECONDARY OUTCOMES:
Occurrence of a low energy vertebral fracture and non vertebral fracture | Baseline, 1 year, 2 years and 3 years
  Lateral and front lumbar x-ray
BMD at the total left hip | Baseline, 3 years
  Dual energy x-ray absorptiometry at lumbar spine (L2-L4)
BMD at lumbar spine and the total left hip | Baseline, 1 year, 2 years
  Dual energy x-ray absorptiometry at left femoral neck and total left hip
Biological assays with bone turnover marker of resorption and tryptase levels to assess mastocytosis activity | Baseline, then every 6 months in 3 years
  Withdrawal of 45 ml of blood
Number of serious adverse events to evaluate drug tolerance | Every 6 months in 3 years
  * Biological assessment: complete blood count, creatinemia, electrolytes, aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin, c-reactive protein (CRP), phosphocalcic analyses with calcemia, phosphoremia, parathormone, vitamin D (25-OH-D), β-Human Chorionic Gonadotropin (HCG) (if needed)
  * Clinical assessment: blood pressure, pulse, weight, height, PS, temperature
Number of non-serious adverse events to evaluate drug tolerance | Every 6 months in 3 years
  * Biological assessment: complete blood count, creatinemia, electrolytes, aspartate aminotransferase (AST), alanine aminotransferase (ALT), bilirubin, c-reactive protein (CRP), phosphocalcic analyses with calcemia, phosphoremia, parathormone, vitamin D (25-OH-D), β-Human Chorionic Gonadotropin (HCG) (if needed)
  * Clinical assessment: blood pressure, pulse, weight, height, PS, temperature
Annual variation of BMD in placebo group and number of low energy fracture compared to historical postmenopausal data | Baseline, 1 year, 2 years, 3 years
  Dual energy x-ray absorptiometry at lumbar spine (L2-L4), left femoral neck and total left hip

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hermine, MD, Study Director — Assistance Publique - Hôpitaux de Paris; Laurent FRENZEL, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (11):
- France (11):
  - Jean Minjoz Hospital, Dermatology department, Besançon
  - Caen Hospital, Clinical haematology department, Caen
  - Estaing Hospital, Cellular therapy and clinical haematology department, Clermont-Ferrand
  - Lille CHRU Hospital, Internal medicine and clinical immunology department, Lille
  - La Timone Hospital, Dermatology and cutaneous oncology department, Marseille
  - Lapeyronie Hospital, Rheumatology and Immunology department, Montpellier
  - La Pitié-Salpêtrière Hospital, Internal medicine and clinical immunology department, Paris
  - Cochin Hospital, Rheumatology department, Paris
  - Necker Hospital, Adult haematology department, Paris
  - Strasbourg Hospital, Rheumatology department, Strasbourg
  - Toulouse Hospital, Dermatology department, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johnson MR, Verstovsek S, Jorgensen JL, Manshouri T, Luthra R, Jones DM, Bueso-Ramos CE, Medeiros LJ, Huh YO. Utility of the World Heath Organization classification criteria for the diagnosis of systemic mastocytosis in bone marrow. Mod Pathol. 2009 Jan;22(1):50-7. doi: 10.1038/modpathol.2008.141. Epub 2008 Sep 19. PMID 19116630
- [Background] Theoharides TC, Valent P, Akin C. Mast Cells, Mastocytosis, and Related Disorders. N Engl J Med. 2015 Jul 9;373(2):163-72. doi: 10.1056/NEJMra1409760. No abstract available. PMID 26154789
- [Background] Frenzel L, Hermine O. Mast cells and inflammation. Joint Bone Spine. 2013 Mar;80(2):141-5. doi: 10.1016/j.jbspin.2012.08.013. Epub 2012 Oct 30. PMID 23116710
- [Background] Rabenhorst A, Christopeit B, Leja S, Gerbaulet A, Kleiner S, Forster A, Raap U, Wickenhauser C, Hartmann K. Serum levels of bone cytokines are increased in indolent systemic mastocytosis associated with osteopenia or osteoporosis. J Allergy Clin Immunol. 2013 Nov;132(5):1234-1237.e7. doi: 10.1016/j.jaci.2013.06.019. Epub 2013 Jul 31. No abstract available. PMID 23910691
- [Background] Barete S, Assous N, de Gennes C, Grandpeix C, Feger F, Palmerini F, Dubreuil P, Arock M, Roux C, Launay JM, Fraitag S, Canioni D, Billemont B, Suarez F, Lanternier F, Lortholary O, Hermine O, Frances C. Systemic mastocytosis and bone involvement in a cohort of 75 patients. Ann Rheum Dis. 2010 Oct;69(10):1838-41. doi: 10.1136/ard.2009.124511. Epub 2010 Jun 22. PMID 20570833
- [Background] van der Veer E, Arends S, van der Hoek S, Versluijs JB, de Monchy JGR, Oude Elberink JNG, van Doormaal JJ. Predictors of new fragility fractures after diagnosis of indolent systemic mastocytosis. J Allergy Clin Immunol. 2014 Dec;134(6):1413-1421. doi: 10.1016/j.jaci.2014.05.003. Epub 2014 Jun 27. PMID 24985401
- [Background] Rossini M, Zanotti R, Viapiana O, Tripi G, Idolazzi L, Biondan M, Orsolini G, Bonadonna P, Adami S, Gatti D. Zoledronic acid in osteoporosis secondary to mastocytosis. Am J Med. 2014 Nov;127(11):1127.e1-1127.e4. doi: 10.1016/j.amjmed.2014.06.015. Epub 2014 Jun 20. PMID 24954632
- [Background] Edwards BJ, Bunta AD, Lane J, Odvina C, Rao DS, Raisch DW, McKoy JM, Omar I, Belknap SM, Garg V, Hahr AJ, Samaras AT, Fisher MJ, West DP, Langman CB, Stern PH. Bisphosphonates and nonhealing femoral fractures: analysis of the FDA Adverse Event Reporting System (FAERS) and international safety efforts: a systematic review from the Research on Adverse Drug Events And Reports (RADAR) project. J Bone Joint Surg Am. 2013 Feb 20;95(4):297-307. doi: 10.2106/JBJS.K.01181. PMID 23426763
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655